CLINICAL TRIAL: NCT06522646
Title: Evaluation of a Microprocessor-controlled Prosthetic Knee-ankle System (SPCM)
Acronym: SPCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institution Nationale des Invalides (Other)
Collaborators: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other); Hopital d'instruction des armées Percy (HIA Percy) (Unknown); Proteor Group (Industry); Direction Générale de l'Armement (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPCM
Record Dates: First submitted 2024-07-16; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Amputation; Lower Limb Amputation Above Knee (Injury)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPCM (Experimental): Patients will be fitted with the SPCM prothesis
  Interventions: Device: SPCM
- Usual Prosthesis (Active Comparator): Patients will be fitted with their usual microprocessor prosthesis
  Interventions: Device: Usual Prothesis

INTERVENTIONS:
Device: SPCM — During a period of 4-6 weeks, patients will live in their usual environment with the SPCM prosthesis
  Arms: SPCM
Device: Usual Prothesis — During a period of 4-6 weeks, patients will live in their usual environment with their usual microprocessor prosthesis
  Arms: Usual Prosthesis

SUMMARY:
The main aim of this study is to compare the adaptation capabilities of the microprocessor-controlled knee-ankle prosthesis system with the comparator covered by the French LPPR, known as the "usual prosthesis".

The main hypothesis being that wearing the SPCM increases the time spent flat-footed in the various walking situations of everyday life, bringing it closer to that of asymptomatic people.

This is a prospective, multicenter, randomized, cross-over study. The participants are transfemoral amputees who have been fitted with a microprocessor-controlled prosthetic knee for more than 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Amputee at or above knee level
* Person fitted for more than 3 months with a microprocessor-controlled knee support phase and oscillating phase, in accordance with the conditions for reimbursement set out in the LPPR.
* Person with a level of activity according to the International Classification of of Functioning, Disability and Health greater than or equal to d4602 (moving around outside the house and other buildings)
* Person able to understand simple commands, to read and write, and to give their informed consent
* Person who has given informed consent
* Person affiliated to a social security scheme

Exclusion Criteria:

* Minor
* Person of full age subject to a legal protection measure or unable to express consent
* Pregnant or breast-feeding women
* Persons with bilateral amputations
* Person with a neurological or orthopedic pathology with major repercussions on locomotion
* Persons with a ground/knee height of less than 43.5 cm or more than 55 cm
* Persons weighing more than 125 kg
* Foot size less than 24 cm or greater than 30 cm
* Person with a hip disarticulation
* Person without an emergency walking solution
* Person with a suspension fitting with vacuum pump
* Person planning a trip outside Europe or unable to return in less than 24 hours (in case of device failure) for the duration of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the time (measured as a percentage of the gait cycle) when the foot is flat on the ground during walking in three gait situations: flat, on a slope and going down stairs, with SPCM and the usual prosthesis. | Evaluation after 4 weeks' wear of each of the 2 prostheses
  The aim is to compare the adaptation of the prosthetic system to the constraints of everyday life. SPCM adapts the ankle's behavior to the walking situation, and should make it possible to restore the time during which the foot remains flat during the stance phase, in different situations

SECONDARY OUTCOMES:
Contralateral ankle power | Evaluation after 4 weeks' wear of each of the 2 prostheses
  Contralateral ankle power is a locomotor compensation device used by transfemoral amputees. It is a biomechanical parameter usually measured by quantified motion analysis (AQM). The SPCM prosthetic system is expected to reduce these power.
Pelvis elevation | Evaluation after 4 weeks' wear of each of the 2 prostheses
  Pelvis elevation is a locomotor compensation device used by transfemoral amputees. It is a biomechanical parameter usually measured by quantified motion analysis (AQM). The SPCM prosthetic system is expected to reduce these Pelvis elevation.
Toe clearance | Evaluation after 4 weeks' wear of each of the 2 prostheses
  Toe clearance is the distance between the toe of the foot and the ground during the swing phase. The greater this distance, the safer the patient. With SPCM, the toe clearance should increase, providing greater safety during pitch change in the swing phase.
Prosthesis evaluation | Evaluation after 4 weeks' wear of each of the 2 prostheses
  The PEQ is composed of 9 validated scales that are each comprised of multiple questions, and there are a number of additional individual questions. Each question is rated between 0 and 100. Higher number will correspond with a more positive response.
Locomotor abilities | Evaluation after 4 weeks' wear of each of the 2 prostheses
  It is composed of 14 questions about different locomotor activities. A 4-level ordinal scale (0-3 points; ranging from "not able" to "able to accomplish the activity alone") scores the degree of a person's perceived independence in performing each of the 14 activities while wearing the prosthesis. The higher the total score, the greater the patient's abilities.
Mobility | Evaluation after 4 weeks' wear of each of the 2 prostheses
  The Prosthetic Limb Users Survey of Mobility (PLUS-M) is a self-report instrument for measuring mobility of adults with lower limb amputation. PLUS-M provide a T-score that ranges from 17.5 to 76.6.A higher PLUS-M™ T-score corresponds to greater mobility.
SF-36 Questionnaire | Evaluation after 4 weeks' wear of each of the 2 prostheses
  Socre of the SF-36 questionnaire, evaluation of the quality of life. The score range from 0 to 100. A higher score mean a better outcome.
Number of steps | Evaluation after 4 weeks' wear of SPCM
  Quantifying real-life activity. The aim is to check whether the improvements observed during the laboratory motion analysis test are reflected in real life.
  Comparison of the number of steps recorded by the prosthesis sensors and those obtained during the laboratory gait analysis. Equivalence between the systems is expected.
Cadence | Evaluation after 4 weeks' wear of SPCM
  Quantifying real-life activity. The aim is to check whether the improvements observed during the laboratory motion analysis test are reflected in real life.
  Comparison of the cadence recorded by the prosthesis sensors and those obtained during the laboratory gait analysis. Equivalence between the systems is expected.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital d'Instruction des Armées (HIA) Percy, Clamart
  - UGECAM-NE - Institut Régional de Médecine Physique et de Readaptation de Nancy, Nancy
  - Insitution Nationale des Invalides, Paris
  - Institut de Biomécanique Humaine Georges Charpak, Paris

IPD SHARING:
Plan to Share IPD: No